CLINICAL TRIAL: NCT06676631
Title: NK010 or NK042 Cell Injection in Combination With Rituximab in Patients With Refractory Systemic Lupus Erythematosus or Lupus Nephritis
Brief Title: NK010 or NK042 in Combination With Rituximab for Refractory Systemic Lupus Erythematosus/Lupus Nephritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK010-NK042-I-SLE-01
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Refractory Systemic Lupus Erythematosus; Refractory Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK 010 or NK 042 infusion (Experimental): Subjects with refractory SLE or LN will receive rituximab followed by NK010 or NK042.
  Interventions: Biological: NK 010 or NK042; Drug: Rituximab

INTERVENTIONS:
Biological: NK 010 or NK042 — NK010 is an allogeneic non-genetically modified NK cell infusion. NKX010 will be administered at a dose of 2.5 × 109 NK cells, 5.0 × 109 NK cells and 7.5 × 109 NK cells by a dose-escalation design and administered IV. N042 is an allogeneic genetic modification of NK cell. NKX042 will be administered at a dose of 6 × 108 NKR positive NK cells, 1.2 × 109 NKR positive NK cells and 2.4 × 109 NKR positive NK cells by a dose-escalation design and administered IV.
  Other Names: NK010 or NK042 infusion
Drug: Rituximab — RTX dose of 1 g administered IV over 60 minutes at the first day of the treatment phase.
  Other Names: RTX

SUMMARY:
This is an investigator-initiated, open-label, single-arm study to determine safety and preliminary efficacy of NK010 or NK042 in combination with rituximab (RTX) for the treatment of patients with refractory systemic lupus erythematosus (SLE) or lupus nephritis (LN) in China.

DETAILED DESCRIPTION:
The study will consist of 3 study periods for each study subject inclusive of screening, treatment and follow-up. During the treatment phase, the subjects will receive 1000 mg of rituximab treatment on day 1, followed by NK010 or NK042 treatment on days 4, 6, and 8, respectively. The subject will be followed at the day 14, day 28, Month 2, Month 3, and every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old, male or female.
* A diagnosis of SLE according to the 2019 EULAR (European League Against Rheumatism)/ACR (American College of Rheumatology).
* Inclusion criteria applicable to the LN subgroup: active type III or IV lupus nephritis (with or without type V) confirmed by renal biopsy according to the 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria. An activity index ≥2 and a chronicity index no more than moderate according to the 2018 RPS Task Force for LN pathologic types and the National Institutes of Health (NIH) Lupus Nephritis Activity and Chronicity Index Score criteria. Urine protein/creatinine ratio (UPCR) ≥ 1.0 g/g or 24-hour urine protein quantification ≥ 1.0 g/day.
* One of the following at screening: positive antinuclear antibody (ANA) OR positive anti-dsDNA OR positive anti-Smith antibody.
* SLEDAI-2000 score ≥ 8.
* Prior to screening, having received glucocorticoids combined with immunosuppressants and/or biologics for at least 3 months with stable doses for >2 weeks, but disease still active (i.e., received glucocorticoids + immunosuppressants or glucocorticoids + immunosuppressants + biologics; monotherapy with any of the above drugs is not eligible).
* Hematologic, hepatic, renal, pulmonary, and cardiac function criteria at screening were as follows: ① leukocytes ≥ 2 ×109/L and lymphocyte count ≥ 0.5 ×109 /L; ② serum ALT and AST ≤ 3 times the upper limit of normal; ③ total bilirubin ≤ 1.5 times the upper limit of normal, with the exception of patients with Gilbert's syndrome, for whom total bilirubin was ≤ 3.0 times the upper limit of normal; ④ eGFR (based on the creatinine based on the CKD-EPI formula) ≥ 30 ml/min/1.73m2; ⑤ oxygen saturation ≥ 92% in non-oxygenated state under indoor ventilation; no clinically significant pleural effusion; ⑥ left ventricular ejection fraction ≥ 45%, and no clinically significant abnormal findings on ECG.
* For participants not receiving therapeutic anticoagulation: International standardized ratio (INR) ≤ 1.5 times the upper limit of normal, or prothrombin time (PT) ≤ 1.5 times the upper limit of normal.
* Participants receiving hematopoietic growth factor support therapy, including erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage-colony-stimulating factor (GM-CSF), and platelet agonists (TPO), must have a 2-week interval between the last growth factor support therapy and the screening period assessment; those receiving blood product transfusion that require at least 1 week between the screening period platelet assessment and the last platelet transfusion, and at least 2 weeks between the screening period hemoglobin assessment and the last red blood cell transfusion.
* Female participants of childbearing potential must have a negative serum pregnancy test at screening (women who are surgically sterilized or have been menopausal for at least 2 years are not considered to be of childbearing potential). Female subjects of childbearing potential and male subjects must use highly effective methods of contraception throughout the clinical study and for 1 year after the last study treatment; they should also commit not to donate eggs (oocytes, oocytes)/sperm for assisted reproduction for 1 year after the last study treatment.
* Participants are willing to participate in this study and sign a paper version of the informed consent form.

Exclusion Criteria:

* Requires dialysis treatment (hemodialysis or peritoneal dialysis) at the time of screening or is expected to require dialysis treatment during study treatment.
* Have received a solid organ or hematopoietic cell transplant or plan to do so during study period.
* Have a congenital or acquired immunodeficiency that results in a serious infection, or are receiving chronic immunoglobulin replacement therapy.
* Presence of active mixed connective tissue or systemic sclerosis, an overlapping syndrome, in the 12 months prior to or during screening, and the adverse condition or other treatment may affect study efficacy or safety assessment or outcomes. Overlapping syndromes in which the anticipated condition or treatment does not affect the assessment or outcome are not excluded.
* Receipt of any B-cell depletion therapy (e.g., anti-CD20, anti-CD19 monoclonal antibody), including but not limited to zolmitriptan in rituximab, obinutuzumab, bortezomib, within 6 months prior to screening; or treatment with any biologic, such as, but not limited to, belimumab, anifrolumab, or tetracycline, within 1 month prior to screening.
* Participants with known anaphylaxis, hypersensitivity, intolerance, or contraindication to NK010 Cell Injection, NK042 Cell Injection, RTX, or any of the components of the drugs that may be used in the study, or subjects who have had a previous severe allergic reaction.
* Clinically significant central nervous system disease or pathological changes not due to lupus within 3 months prior to the first dose, including, but not limited to, cerebrovascular accident (ischemia/hemorrhage), aneurysm, epilepsy, convulsions/convulsions, aphasia, severe brain injury, dementia, parkinson's disease, cerebellar disorders, organic brain syndromes, or psychiatric disorders.
* Unstable cardiovascular function: ① Uncontrollable angina pectoris or life-threatening unstable arrhythmia; ② Myocardial infarction or unstable angina pectoris within 3 months prior to the screening; ③ Previous coronary artery or graft revascularization; ④ Uncontrolled, clinically significant arrhythmia (e.g., sustained ventricular tachycardia, ventricular fibrillation, tip-twisting); ⑤ Mobitz type II Mobitz type II or III atrioventricular block; (6) congestive heart failure or severe cardiac insufficiency with New York Heart Association classification ≥ grade 3; (7) prolongation of the QT interval (QTc) corrected for heart rate (Fridericia) by > 480 milliseconds; (8) uncontrolled hypertension (systolic blood pressure >160 mm Hg and/or diastolic blood pressure > 100 mm Hg), or associated with hypertensive crisis or hypertensive encephalopathy.
* Active bleeding.
* Any active infection, excluding fungal infections of the nail beds; history of severe recurrent or chronic infections.
* Presence of active infection treated with intravenous antibiotics within 14 days prior to screening, except for antibiotic prophylaxis (including intravenous administration).
* Positive serum HIV viral antibodies or history of active HIV infection and positive syphilis antibodies at screening.
* Positive Hepatitis B Surface Antigen (HBsAg). Participants who are HBsAg negative and Hepatitis B Core Antibody (HBcAb) positive, but Hepatitis B Virus (HBV) DNA negative are eligible for enrollment, but will require monitoring of HBV DNA at each follow-up visit.
* Positive Hepatitis C Serology. Participants with hepatitis C antibodies positive but do not have detectable hepatitis C virus (HCV) RNA for at least 6 months after completion of antiviral therapy are eligible for enrollment, but require monitoring of HCV RNA at each follow-up visit.
* Risk of active tuberculosis at screening, with or without completion of adequate treatment, including the presence of signs or symptoms of active tuberculosis (e.g., fever, cough, night sweats, and weight loss) as judged by the investigator at screening; documented active tuberculosis on chest imaging (e.g., chest x-ray, chest CT scan) performed at screening or at any time during the 6 months prior to screening; latent tuberculosis at screening evidence of infection such as a positive gamma-interferon release test.
* Participants with a malignant tumor, including tumor-associated polymyositis/dermatomyositis, within 5 years prior to screening. Except for surgically resected and cured non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, low-stage bladder cancer, ductal carcinoma in situ of the breast, or cured participants with no evidence of recurrence within the last 2 years and no need for treatment.
* Previous received cell therapy such as CAR-T, CAR-NK, ect.
* Pregnant or lactating women, or (if of childbearing potential) subjects who are not using adequate contraception or planning to donate oocytes and sperm.
* The presence of any life-threatening disease, medical condition, or organ system dysfunction that, in the opinion of the Investigator, may affect the safety of the subject or compliance with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate for SLE response index 4 (SRI4) | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  SRI4 response defined as a reduction of ≥4 points on SLEDAI-2000, no new domain A scores and no more than 1 new domain B score on BILAG 2004, and no deterioration in PGA (<0.3 point increase).
Number of participants who achieved renal response | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  For subjects with LN: evaluate the number of participants achieved complete renal response (CRR) and partial renal response (PRR) according to European Alliance of Associations for Rheumatology (EULAR)/European Renal Association-European Dialysis and Transplantation Association (ERA-EDTA) criteria.
Number of subjects who achieved lupus low disease activity state (LLDAS) | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  Low lupus disease activity was defined as (i) SLEDAI-2K total score ≤ 4, no active lesions in major organ systems (including kidney, central nervous system, cardiopulmonary, vasculitis, and fever) and no hemolytic anemia or gastrointestinal lesions; (ii) no new indications of lupus disease activity compared with previous evaluations (according to SLEDAI-2K); (iii) Physician's Global Assessment (PGA) ≤ 1; and (iv) prednisone ≤ 7.5 mg d for use of malaria and biologic agents. Assessment (PGA) ≤ 1 point; ④ Prednisone ≤ 7.5 mg/d, maintenance of standard therapy. biologics.
Number of participants who achieved clinical remission of SLE | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  Clinical remission of SLE was defined by 2021 DORIS SLE remission criteria.
The change of Physician Global Assessment (PGA) score | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  The change of PGA score will be compared to baseline.
The change of SLEDAI-2000 scores | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  The change of SLEDAI-2000 score will be compared to baseline.
Changes of autoantibody of SLE from baseline | Day 14, day 28, 2 months, 3 months, 6 months, 9 months, 12 months after the first administration of NK010 or NK042 infusion
  Autoantibody include anti-dsDNA, anti-nuclear antibody, ANA, anti-Sm antibody, and complement C3, C4.
Dose-limiting toxicity (DLT) rate | 28 days after initial study treatment.
  This is to measure the dose-limiting toxicity of NK 010 or NK 042.
Incidence of treatment-related adverse events | 1 year
  This is to measure safety and tolerability of NK 010 or NK 042.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdomg, China

IPD SHARING:
Plan to Share IPD: No